CLINICAL TRIAL: NCT06155474
Title: Effects of Prebiotics on Metagenomic Diversity and Abundance in Young Children With Acute Malnutrition: A Double-blinded Randomised Controlled Trial (PMAM)
Brief Title: Effects of Prebiotics on Metagenomic Diversity and Abundance in Young Children With Acute Malnutrition
Acronym: P-MAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of the Punjab (Other)
Collaborators: University of Veterinary and Animal Sciences, Lahore - Pakistan (Other)
Responsible Party: Principal Investigator, Dr. Javeria Saleem, Assistant Professor, University of the Punjab
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D/137/FIMS
Record Dates: First submitted 2023-10-17; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Child Malnutrition
Keywords: malnutrition; Metagenomics; Micro-biota
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition | interventions — Powders; Starch

STUDY DESIGN:
Intervention Model Description: Prebiotic
Who Masked: Participant, Investigator
Masking Description: During trial conduct, the following groups will all be blinded to participants' allocation Healthy/Control, Malnutrition (RUTF) and Malnutrition (RTUF + prebiotics)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy/Control (Starch) (Placebo Comparator): The Healthy Controls will be given starch packed in the same way as the active prebiotics
  Interventions: Dietary Supplement: Starch Only
- Malnutrition (RUTF + Starch) (Experimental): The Malnutrition group with RUTF and Starch only. The RUTF will be given as per the WHO guidelines
  Interventions: Dietary Supplement: RUTF + Starch
- Malnutrition (RUTF + prebiotics) (Active Comparator): The Malnutrition group with RUTF and Prebiotic only. The RUTF will be given as per the WHO guidelines
  Interventions: Dietary Supplement: Prebiotic galacto-oligosaccharide (GOS) Powder

INTERVENTIONS:
Dietary Supplement: Prebiotic galacto-oligosaccharide (GOS) Powder — Prebiotic GOS Powder is a galacto-oligosaccharide ingredient low in mono-sugars. Scientific studies have shown positive effects of oligosaccharides, among which galacto-oligosaccharides, on growth of bifidobacterial, stool consistency bowel function and transit time, support of natural defenses and mineral absorption.
  The product mainly consists of 97% dry matter with 69% prebiotic GOS, 23% lactose and 5% glucose and galactose as monosaccharides. These prebiotics have β-(4) glycosidic linkages and have been proven as safe product
  Arms: Malnutrition (RUTF + prebiotics)
Dietary Supplement: Starch Only — The Starch Solution is a low-fat diet.
  Arms: Healthy/Control (Starch)
Dietary Supplement: RUTF + Starch — ready-to-use therapeutic food and The Starch Solution is a low-fat diet.
  Arms: Malnutrition (RUTF + Starch)

SUMMARY:
Malnutrition is a major global public health issue, contributing to poor health and early morbidities in children under five, particularly in developing countries. In 2021, 5 million children died worldwide due to infectious diseases or malnutrition, with Pakistan having the highest under-five mortality rate. With a population of approximately 229 million, Pakistan is the fifth most populous country in the world. In Pakistan, under-five mortality is 63.3 per 1000 live births which has declined from 139.8 in 1990 to 63.3 in 2021 (WHO, 2022, UNICEF, 2023). The monsoon season's massive flooding in Pakistan has worsened the humanitarian situation, endangering the already vulnerable population. UNICEF reports high rates of acute malnutrition, political instability, economic decline, and coronavirus disease 2019 effects. However, there is limited evidence on the efficacy of probiotics for infants in Pakistan.

Metagenomics is the study of microorganisms' genomes, examining all microorganisms in an ecological site's genomes. It involves extracting and sequencing DNA using high-throughput techniques. Scientists can identify genes with significant features using computer analysis. The distal intestine contains around one trillion organisms per milliliter of luminal contents, and understanding their potential for energy and nutrient harvest is crucial in malnourished individuals.

Alpha diversity is the analysis of species diversity in a sample, measured by observed species index, Chao1 index, Shannon index, Simpson index, and good-coverage index. It is proportional to the first four values and indicates less undiscovered species. The distal intestine contains around one trillion organisms per milliliter of luminal contents, with an increased capacity for energy harvest in malnourished individuals.

The present study aims to measure the following objectives. i. -To estimate the microbiome degree of diversity among malnutrition children micro-biota defined by 16 Svedberg (S) ribosomal ribonucleic acid gene sequencing.

ii. -To evaluate the interpersonal differences in the structure and functioning of the gut microbiome that affect a person's vulnerability to malnutrition.

iii. -To determine how microbiomes are shaped by host genotypes, environmental exposures, including exposure to malnutrition in children mothers, and other family members, nutritional status, and lifestyles, including diet.

DETAILED DESCRIPTION:
Metagenomics is the study of microorganisms' genomes through the direct extraction and cloning of their DNA from a collection of microorganisms, also known as environmental and community genomics. The examination of all the microorganisms in an ecological site's genomes, the majority of which cannot be produced under standard laboratory conditions, is called metagenomics. In order to achieve this, the site's microbial population must first be removed, and then its DNA must be isolated and sequenced using high-throughput techniques. Scientists may identify genes with significant features, such as virulence genes or genes encoding enzymes of commercial significance, using computer analysis of a sequence.

Around one trillion organisms per milliliter of luminal contents are found in the distal intestine, where the majority of these bacteria are found. It is essential to describe the microbiota and its microbiome in malnourished persons and to define their potential to harvest energy and nutrients in light of the discovery that the intestinal microbiota/ microbiome linked with obesity has an increased capacity for energy harvest.

Deficiency of iron has been recognized in malnourished children. Iron present in RUTF is not sufficient to elevate "circulating levels of ferritin into the optimal physiological range. Prebiotics has been proven to have anti-inflammatory and antimicrobial actions that might enhance response to standard therapy for severe acute malnutrition (SAM), Targeting the gut microbiota through the use of Prebiotics as part of treatment in malnourished children may present an affordable and cost-effective strategy in the prevention and also in the treatment Fortifying the microbiota with Prebiotics could enhance energy and may protect against diarrhoea. However, randomized controlled trials evaluating the effects of prebiotic supplementation in children with severe acute malnutrition have not previously been done. So clinical evidence is lacking and cannot be translated into clinical practice.

Content of "Ready-to-use therapeutic food" may not be optimal to support weight gain a in children with severe acute malnutrition. Further trials are required to conclude whether Prebiotics containing Galactooligosaccharides supplement can improve weight gain in children with severe acute malnutrition in other settings.

Trial Objectives and Endpoints Trial Objectives

* To estimate the microbiome degree of diversity among malnutrition children micro-biota defined by 16 Svedberg (S) ribosomal ribonucleic acid gene sequencing.
* To evaluate the interpersonal differences in the structure and functioning of the gut microbiome that affect a person's vulnerability to malnutrition.
* To determine how microbiomes are shaped by host genotypes, environmental exposures, including exposure to malnutrition in children mothers, and other family members, nutritional status, and lifestyles, including diet.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria: Age 6-59 months at enrolment;
* Acute malnutrition without complications, as defined by the World Health Organization (i.e., children with mid-upper arm circumference (MUAC) <115 mm or weight-for-height z-score <-3 or grade 1-2 bilateral edema who will be clinically well and alert with good appetite);
* Parental consent for the child to participate.
* Healthy children without any chronic or acute illness

Exclusion Criteria:

* Presence of any complications of severe malnutrition (severe dehydration, severe anemia, severe pitting edema, anorexia, hypothermia, high pyrexia, acute lower respiratory infection, or hypoglycemia) or immunocompromised.
* Children on antibiotic treatment for any disease in the last 3 months will be excluded.

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Microbiome diversity | 8 Weeks
  Microbiome diversity examination among malnourished children using 16 Svedberg (S) ribosomal ribonucleic acid gene sequencing. The microbiome diversity index measures the diversity of microbial species in malnourished children's gut microbiota, comparing it to reference or control populations. Higher values indicate greater diversity, providing insights into malnutrition's impact on gut microbiota composition.

SECONDARY OUTCOMES:
Anthropometric Measurements | 8 Weeks
  Change in the mean weight-for-height/length z-score in children with complicated severe acute malnutrition who have been taking prebiotics supplementation for 8 weeks.
Neurodevelopment Assessment | 8 Weeks
  Impact assessment of prebiotic supplementation on children's neurodevelopment using the Malawi Development Assessment tool
Muscle mass accumulation | 8 Weeks
  The study investigates the impact of prebiotic consumption on body composition changes using the Body Stat Analyzer as a quantitative measurement tool.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Public Health, University of the Punjab, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saleem J, Zakar R, Iqbal S, Arshad M, Shahzad R, Batool M, Nawaz M, Butt MS, Fischer F. Effects of prebiotics on microbial diversity and abundance in young children with acute malnutrition: study protocol for a multi-centered, double-blinded randomized controlled trial. Trials. 2024 Nov 26;25(1):798. doi: 10.1186/s13063-024-08647-z. PMID 39593072